CLINICAL TRIAL: NCT01052064
Title: Therapy With rTMS in Children With Attention Deficit and Hyperactivity Disorder. Phase 1 Study.
Brief Title: Transcranial Magnetic Stimulation in Children With Attention Deficit Hyperactivity Disorder (ADHD). A Safety Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Center for Neurological Restoration, Cuba (Other)
Responsible Party: Lázaro Gómez Fernández, MD, International Center for Neurological Restoration
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rTMS-09.01-ADHD
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Children; ADHD; rTMS; Safety
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcranial magnetic stimulation (Experimental): There are evidences that rTMS has a modulating effect in cortical and subcortical neural networks, reinforcing or depressing synaptic activity by mean of long term potentiation or depression like mechanism. Depression is the most study neuropsychiatric condition in which rTMS is useful as a therapeutic option; but in other diseases such as ADHD there are many pathophysiological elements that make it very likely that rTMS could be useful for symptomatic treatment modulating activity in prefrontal and basal ganglia neuronal networks.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — rTMS will be administered in one daily session during 5 consecutive days of 1 Hz, 90% of motor threshold for a total of 1500 stimuli. The stimulation will be focal over left dorsolateral-prefrontal cortex(F3, from the international 10-20 system)
  Other Names: Repetitive Transcranial Magnetic Stimulation(rTMS)

SUMMARY:
Low frequency repetitive Transcranial Magnetic Stimulation(rTMS) is a safe and tolerable procedure in children with Attention Deficit Hyperactivity Disorder(ADHD); it also could be a complement to the treatment of patients with poor symptomatic control to conventional treatment.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder is a common disorder in the infancy; the majority of ADHD have good clinical response to amphetamines alone or in association with antiepileptic drugs. It is described that some patients(10-30%) with ADHD do not respond to conventional pharmacological and psycho- pedagogical treatment; in those patients non invasive brain stimulation methods could be a supplementary option for symptomatic control. There are not many published papers describing the effects of rTMS in persons younger than 18 years; so the first step to extent its use in pediatric population should be to obtain evidences about its tolerance and safety.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for Study: 7years to 12 years
* Genders Eligible for Study: Both

Exclusion Criteria:

* History of convulsions
* Co-morbidity with other psychiatric or neurologic disease

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | week 1,during treatment

SECONDARY OUTCOMES:
EEG changes in epileptiform or basal activity after treatment compared with the baseline | last day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lázaro Gómez, MD, Principal Investigator — International Center of Neurological Restoration
Locations (1):
- International Center for Neurological Restoration, Havana, La Habana, Cuba